CLINICAL TRIAL: NCT07000708
Title: VITAL: Vaccination, Immunity, Time-restricted Eating, Aging and Lifestyle
Acronym: VITAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Max Delbrück Center for Molecular Medicine (MDC), Berlin (Unknown); Labor Berlin, Germany (Unknown); Experimental & Clinical Research Center Berlin (Unknown); University of Oxford (Other); University of Cologne (Other)
Responsible Party: Principal Investigator, Sebastian Hofer, Dr. rer. nat., Dr. rer. nat., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EA4/154/24
Record Dates: First submitted 2025-04-30; First posted 2025-06-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Vaccination; Immunosenescence; Metabolism
Keywords: fasting; vaccination; intermittent fasting; time-restricted eating; influenza; immunity; aging; immunosenescence
MeSH Terms: conditions — Fasting; Intermittent Fasting; Influenza, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (no intervention) (No Intervention): Four weeks of ad libitum eating pattern with eating time window >11 h/day. No change of the regular eating pattern.
- TRE (Experimental): Four weeks of TRE, where the daily eating pattern is reduced to 8 h/day. The first meal will be before 10:00 AM.
  Interventions: Behavioral: TRE: Time-restricted eating

INTERVENTIONS:
Behavioral: TRE: Time-restricted eating — The daily eating pattern is reduced to 8 h/day. The first meal will be before 10:00 AM.
  Arms: TRE

SUMMARY:
The aim of this study is to investigate the effects of a four-week time-restricted eating (TRE) intervention on autophagy, immune function, and vaccine response to a seasonal influenza and COVID-19 vaccines in older healthy subjects.

DETAILED DESCRIPTION:
Aging impairs immune cell autophagy and reduces vaccine efficacy, leaving older adults highly vulnerable to influenza and other infectious diseases. Time-Restricted Eating (TRE), by limiting daily food intake to an 8-hour window without detailed calorie counting, modulates nutrient-sensing pathways (e.g., mTOR inhibition, AMPK activation) and boosts autophagic flux in preclinical models. In a randomized, controlled trial, healthy volunteers aged 60-85 will follow either four weeks of TRE or their usual eating pattern. After that, all will receive a standard seasonal vaccines against influenza and COVID-19 outside of the trial at their general practitioner (min. 2 days and max. 14 days after the stop of intervention). Blood and physiologic measurements at baseline, after four weeks of study intervention will quantify autophagy in immune cells, metabolome/proteome shifts, body composition, blood pressure, and arterial stiffness, among others. At two additional visits after the vaccination (2 weeks and 12-14 weeks after the vaccination), immune responses to the vaccination will be monitored in the blood. The investigators hypothesize that TRE-induced restoration of autophagy and amelioration of immunosenescence will correlate with stronger vaccine responses, offering a simple, low-cost strategy to rejuvenate immunity and improve preventive care in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, enrolled in a 1:1 ratio
* Age 60-85 years
* Body mass index (BMI) 20-35 kg/m²
* Capacity to give informed consent
* Existing health insurance to allow evaluation and treatment of any incidental findings
* Usual daily eating window > 11 hours
* First meal of the day before 10:00 AM
* Willingness to receive seasonal influenza and COVID-19 vaccination and proof of scheduled appointment
* Willingness and ability to follow a prescribed TRE dietary regimen (8-hour daily eating window; 16-hour fast without any caloric intake)
* Appointment for simultaneous influenza and COVID-19 vaccination pre-arranged with primary care physician and coordinated with study team to align with TRE intervention

Exclusion Criteria:

* Any vaccination (especially influenza and/or COVID-19) within 6 months before the intervention start
* Vaccinations not related to the study, administered during the study period from V0 to V4
* History of influenza infection within 6 months prior to initiation of the study intervention
* History of severe adverse reactions to prior vaccinations
* Use of pharmacological weight-loss agents (e.g., semaglutide)
* Diabetes mellitus under ongoing pharmacological treatment
* Symptoms of systemic inflammatory or autoimmune disease
* Immunosuppression (including use of immunosuppressive drugs)
* Severe hypertension (systolic > 180 mmHg or diastolic > 110 mmHg)
* Diseases or functional disorders which, in the opinion of the study physician, preclude participation in the study
* Participation in any fasting intervention (e.g., TRE, alternate-day fasting, 5:2, 18:6) within 6 months before enrollment
* Participation in another diet or weight-loss program (e.g., intensive athletic training)
* Night-shift or rotating-shift work
* Severe, active, or unstable medical conditions requiring treatment
* Postoperative recovery phase
* Antibiotic therapy within 3 months before enrollment
* Acute or chronic infections
* Therapeutic or medically prescribed special diets
* Vegan diet
* Current smoker
* Weight change > 2 kg in the month before enrollment
* Known substance, drug, or alcohol abuse
* Anemia
* Claustrophobia
* Legal incapacity or any other circumstance that prevents full understanding of the nature, importance, and implications of the study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Autophagic flux in PBMCs | Change from baseline to 4 weeks
  Change in autophagic flux in peripheral immune cells from baseline (V1) to four weeks (V2), comparing the TRE group versus control, as measured by flow cytometry detection of LC3-II accumulation via antibody staining.

SECONDARY OUTCOMES:
Change in body weight | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in body weight
Change in body composition (BodPod) | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in body composition (e.g., fat and lean body mass), assessed via Air Displacement Plethysmography (ADP, BodPod).
Change in body composition (BIA) | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in body composition (e.g., fat and lean body mass), assessed via bioimpedance analysis (BIA).
Change in the differential blood count | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in the differential blood count, assessed with Hematology analyzers.
Change in blood glucose levels | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in blood glucose levels, assessed via routine blood diagnostic tests
Change in insulin metabolism | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Changes in insulin metabolism parameters, including insulin, IGF-1, C-peptide, ghrelin, leptin, adiponectin, and glucagon, assessed via ELISAs
Changes in blood ketone body levels | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Changes in blood ketone body levels (3-hydroxybutyrate, acetoacetate, acetone), assessed using commercially available assay kits
Change in blood lipid profile | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Changes in blood lipids assessed via metabolomics and routine blood diagnostic tests
Change in liver or renal function | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Changes in blood parameters of liver and renal function assessed via routine blood diagnostic tests
Change in blood electrolyte levels | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Changes in blood electrolyte levels assessed via routine blood diagnostic tests
Change in the incidence of clinically diagnosable infections during the study period | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in the incidence of clinically diagnosable infections during the study period, assessed at study visits by the study physician
Change in continuous blood glucose levels | CGMs will be applied at V1 and V2 and record continuous glucose levels for 14 days each.
  Change in continuous blood glucose levels, assessed with continuous glucose monitors (CGM). CGMs will be applied at V1 and V2 and record continuous glucose levels for 14 days each.
Change in grip strength | Change from baseline to 4 weeks (end of TRE).
  Change in grip strength, assessed with a dynamometer. Handgrip strength will be measured using a dynamometer three times sequentially and repeated after 1 hour.
Change in metabolic rate | Change from baseline to 4 weeks (end of TRE).
  Change in metabolic rate via indirect calorimetry. Indirect calorimetry will be performed to assess energy expenditure as well as carbohydrate and fat oxidation rates. During the procedure, the subject will rest quietly in bed while wearing a ventilated hood. The hood is equipped with an inlet and an outlet valve. Through the inlet valve, the subject receives a constant supply of fresh air, while exhaled air is collected via the outlet valve. Sampling at the rear of the calorimetry device allows determination of gas concentrations in the ambient room air. By calculating the difference, oxygen consumption (VO₂) and carbon dioxide production (VCO₂) in ml/min are determined. These volumes enable the calculation of energy expenditure and substrate oxidation rates. This measurement is performed after a rest period of 30 minutes to determine resting fasting energy expenditure (duration approximately 30 minutes).
Change in Sleep Quality | Change from baseline to 4 weeks (end of TRE)
  Change in Sleep Quality assessed using a questionnaire for the Pittsburgh Sleep Quality Index [PSQI].
Change in health-related quality of life | Change from baseline to 4 weeks (end of TRE)
  Change in EQ-5D-5L assessed using questionnaires.
Change in ChronoType | Change from baseline to 4 weeks (end of TRE)
  Change in ChronoType assessed using the Munich ChronoType Questionnaire [MCTQ]
Change in the Multidimensional Prognostic Index (MPI). | Change from baseline to 4 weeks
  Change in the MPI for geriatric assessment. MPI assessments will be conducted, including documentation of medication and dietary supplement use, medication allergies, nutritional therapies, a range of disease symptoms, social history, activities of daily living (ADL), instrumental activities of daily living (IADL), malnutrition screening, the Short Portable Mental Status Questionnaire (SPMSQ), and the Exton Smith Scale (assessment of decubitus risk), all administered via standardized questionnaires.
Change in the walking speed. | Change from baseline to 4 weeks
  A 10-meter walk test will be performed to determine walking speed in m/s. For this purpose, the subject will walk from a 0-meter mark to a 10-meter mark upon command. Timing will begin at the 2-meter mark. The procedure will be repeated three times, and the times will be averaged. If the subject's fitness level permits, the procedure will be repeated with the instruction to complete the 10 meters 'as fast as possible while still feeling safe'.
Change in proteome profiles in plasma and PBMCs. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in proteome profiles in plasma and PBMCs, measured by LC-MS mass spectrometry or Olink proteomics.
Change in metabolite patterns in plasma. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in metabolite patterns in plasma, assessed by untargeted (¹H-NMR) and/or targeted (LC-MS) metabolomics.
Change in metabolite patterns in stool. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in metabolite patterns in stool, assessed by untargeted (¹H-NMR) and/or targeted (LC-MS) metabolomics.
Change in metabolite patterns in urine. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in metabolite patterns in urine, assessed by untargeted (¹H-NMR) and/or targeted (LC-MS) metabolomics.
Change in gut microbiome composition. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in gut microbiome composition by metagenomic sequencing of stool.
Change in immune-cell subset distribution and activation. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in immune-cell subset distribution and activation, assessed by scRNA-seq and flow cytometry.
Change in body fat percentage. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in body fat percentage, measured by air-displacement plethysmography.
Change in office systolic and diastolic blood pressure. | Change from baseline to 4 weeks
  Change in office systolic and diastolic blood pressure (mmHg), measured by non-invasive blood pressure cuff.
Change in pulse-wave velocity. | Change from baseline to 4 weeks
  Change in pulse-wave velocity (m/s), measured by PulsePen.
Change in frequency of pro- and anti-inflammatory immune cells. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in frequency of pro- and anti-inflammatory immune cells in PBMCs, by flow cytometric immunophenotyping.
Change in immune-cell function. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in immune-cell function (cytokine production, proliferation) after in vitro stimulation of PBMC subsets, by flow cytometry.
Change in circulating pro- and anti-inflammatory cytokine concentrations in plasma. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in circulating pro- and anti-inflammatory cytokine concentrations in plasma, by multiplex cytokine assay.
Change in expression of senescence markers in immune-cell subsets. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in expression of senescence markers in immune-cell subsets, by flow cytometry.
Change in the hypusination status of eIF5A in PBMCs | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in the hypusination status of eIF5A in PBMCs by flow cytometry.
Change in mTOR activity status in PBMCs | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in mTOR activity status in PBMCs by flow cytometry.
Change in expression of key autophagy-regulatory genes. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in expression of key autophagy-regulatory genes in specific immune-cell types or bulk PBMCs, by qPCR, scRNA-seq, or bulk RNA-seq.
Change in energy metabolism in immune-cell subsets. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in cellular energy metabolism in immune-cell subsets, measured by Seahorse extracellular flux analysis and/or Scenith Assay in isolated immune cells ex vivo.
Change in coagulation. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in coagulation, assessed via e.g., thrombin generation, d-dimers from plasma
Change in influenza-specific B- and T-cell responses. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in influenza-specific B- and T-cell responses in serum and PBMCs (e.g., ELISpot).
Change in SARS-CoV-2 specific B- and T-cell responses. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in SARS-CoV-2 specific B- and T-cell responses in serum and PBMCs (e.g., ELISpot).
Change in concentration of influenza-specific IgG antibodies. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in concentration of influenza-specific IgG antibodies, by ELISA.
Change in concentration of SARS-CoV-2 specific IgG antibodies. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in concentration of SARS-CoV-2 specific IgG antibodies, by ELISA.
Change in concentration of influenza-neutralizing antibodies. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in concentration of influenza-neutralizing antibodies.
Change in concentration of SARS-CoV-2 neutralizing antibodies. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in concentration of SARS-CoV-2 neutralizing antibodies.
Change in DNA-break profiles in primary B cells. | Change from baseline to 4 weeks (end of TRE), 2 weeks and 12-14 weeks after vaccination
  Change in DNA-break profiles in primary B cells, assessed by SWIBRID (Switch-joint Breakpoint Repertoire Identification).

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Hofer, Dr. rer. nat., Principal Investigator — Clinical Research Unit, Experimental and Clinical Research Center, Charité, Berlin, Germany & Max-Delbrück Center for Molecular Medicine, Berlin, Germany; Anna Katharina Simon, Prof. Dr., Principal Investigator — Max-Delbrück Center for Molecular Medicine, Berlin, Germany
Locations (1):
- Clinical Research Unit, Experimental & Clinical Research Center, Campus Buch, Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically and scientifically sound proposal.